CLINICAL TRIAL: NCT02435043
Title: A Randomized Controlled Trial of Nature-based Post-stroke Fatigue Rehabilitation (NASTRU)
Brief Title: A Trial of Nature-based Post-stroke Fatigue Rehabilitation (NASTRU)
Acronym: NASTRU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other); Swedish University of Agricultural Sciences (Other); Epidemiology and Register Centre South (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012/352
Record Dates: First submitted 2015-04-07; First posted 2015-05-06 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nature based rehabilitation (Experimental): ten weeks of nature-based rehabilitation, as add-on to standard management
  Interventions: Other: Nature based rehabilitation
- Treatment as usual (Active Comparator): standard management after stroke
  Interventions: Other: standard management after stroke

INTERVENTIONS:
Other: Nature based rehabilitation — ten weeks of nature-based rehabilitation, as add-on to standard management. A rehabilitation program in groups up to 8 patients in an especially designed garden at the Swedish University of Agricultural Sciences, Alnarp. The intervention was grounded in environmental psychology and occupational therapy, supported by a multimodal rehabilitation team that utilized the garden/nature for sensory stimulation, body awareness, meaningful occupations and nature experiences.
  Arms: Nature based rehabilitation
Other: standard management after stroke — standard management after stroke is individualised.
  Arms: Treatment as usual

SUMMARY:
The aim of NASTRU was to examine whether ten weeks of nature-based rehabilitation, as add-on to standard management, could influence post-stroke fatigue (primary outcome), depression, work ability or functional outcome (secondary outcomes), compared to controls.

DETAILED DESCRIPTION:
Patients randomized to the intervention undergo a rehabilitation program in groups up to 8 patients in an especially designed garden at the Swedish University of Agricultural Sciences, Alnarp. The intervention is grounded in environmental psychology and occupational therapy, supported by a multimodal rehabilitation team that utilizes the garden/nature for sensory stimulation, body awareness, meaningful occupations and nature experiences.

The enrollment of 101 patients (51 intervention; 50 control) was completed on August 2014. Follow-up is on-going, with assessments by examiner blinded to treatment group, at end of intervention period, 8 months, and 14 months after randomization. A parallel study with qualitative in-depth interviews in a subset of patients, who were randomized to the intervention group, as well as the staff, is also ongoing.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic or haemorrhagic stroke
* First ever or recurrence, about 3 months (group 1) or more than one year prior to screening (group 2)
* Age: 55-80 years

Exclusion criteria:

* Dementia
* Severe communication disorder that made it difficult to participate and/or serious illnesses besides stroke (for example, serious cancer disease)

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2012-08; Primary Completion 2015-05 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Post stroke fatigue | 8 months after inclusion
  Mental Fatigue Scale (MFS) pre-post design by blinded assessor.
Occupational value of everyday occupation | 8 months after inclusion
  Occupational Value (OVal-pd) pre-post design by blinded assessor

CONTACTS AND LOCATIONS:
Overall Officials: Hélène Pessah-Rasmussen, MD, Ph.D., Principal Investigator — Skane University Hospital
Locations (1):
- Skåne university hospital, Malmo, Sweden